CLINICAL TRIAL: NCT02101372
Title: Gene and Environment in Schizophrenia- Research Groups in Madrid
Brief Title: Intervention Module AGES
Acronym: AGES-CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celso Arango (Other)
Collaborators: Comunidad de Madrid (Other)
Responsible Party: Sponsor-Investigator, Celso Arango, Head of Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2010/BMD-2422
Record Dates: First submitted 2014-03-18; First posted 2014-04-02 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Psychosis
Keywords: first episode psychosis; psychoeducation; group therapy
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment as usual (Active Comparator)
  Interventions: Behavioral: treatment as usual
- Psychoeducation Group (Experimental)
  Interventions: Behavioral: Psychoeducation group treatment

INTERVENTIONS:
Behavioral: treatment as usual — case management
  Arms: treatment as usual
Behavioral: Psychoeducation group treatment — Psychoeducation therapy problem solving focus
  Arms: Psychoeducation Group

SUMMARY:
The AGES-CM consortium aims to study the interaction between the polymorphisms of the candidate genes related with neurodevelopment, neurotransmission, brain progressive changes, cognitive functioning and stressful life events (prospective- and retrospectively assessed) and the association of the interactions with structural and functional brain measures, neuropsychological performance, biochemical and oxidative status in both in patients and controls. The investigators study aimed to examine the effectiveness of a parallel, structured, and specific psychoeducational group intervention (PE) for adolescent patients and their families by comparing it with treatment as usual).

DETAILED DESCRIPTION:
Objective: To assess the effectiveness of a structured psychoeducational group intervention for adolescents with early onset psychosis and their families. The intervention was implemented in parallel in 2 separate groups, by focusing specifically on problem solving strategies and structured psychosis-related information to manage daily life hassles associated with the disease in order to manage crises and prevent relapses.

Method: The investigators performed a 9-month, randomized, rater-blind clinical trial involving adolescent patients with early onset psychosis and 1 or both of their parents. The primary outcomes were number of hospitalizations, days of hospitalization, and visits to the emergency department. The secondary outcome measures were clinical variables and family environment and well being.

ELIGIBILITY:
Inclusion Criteria:

* The presence of at least one positive psychotic symptom (delusions or hallucinations)
* Before age 18 diagnosed by DSM-IV
* Aged between 14 and 19 years and lived at home with 1 or both parents, caregivers, or legal guardians.

Exclusion Criteria:

* The exclusion criteria were patient's drug abuse or dependence at the time of the intervention (drug use was not an exclusion criterion), the presence of any neurological developmental disorder or mental retardation and inability to engage in conversation or read in Spanish that may interfere with the progress of group treatment.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
number of relapses | Change from baseline to 1 -year follow-up and 2 years follow-up

SECONDARY OUTCOMES:
clinical severity | 1year 2 years
  PANSS, CGAS, GAF, CGI-I

CONTACTS AND LOCATIONS:
Overall Officials: Celso Arango, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital general Universitario Gregorio Marañón, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Calvo A, Moreno M, Ruiz-Sancho A, Rapado-Castro M, Moreno C, Sanchez-Gutierrez T, Arango C, Mayoral M. Psychoeducational Group Intervention for Adolescents With Psychosis and Their Families: A Two-Year Follow-Up. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):984-90. doi: 10.1016/j.jaac.2015.09.018. Epub 2015 Oct 13. PMID 26598473
- [Derived] Calvo A, Moreno M, Ruiz-Sancho A, Rapado-Castro M, Moreno C, Sanchez-Gutierrez T, Arango C, Mayoral M. Intervention for adolescents with early-onset psychosis and their families: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):688-96. doi: 10.1016/j.jaac.2014.04.004. Epub 2014 Apr 18. PMID 24839887